CLINICAL TRIAL: NCT00314366
Title: Phase IB Randomized Controlled Double-Blind Trial of Intramyocardial Injection of Autologous Aldehyde Dehydrogenase-Bright Stem Cells Under Electromechanical Guidance for Therapeutic Angiogenesis
Brief Title: Intramyocardial Injection of Autologous Aldehyde Dehydrogenase-Bright Stem Cells for Therapeutic Angiogenesis (FOCUS Br)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Texas Heart Institute (Other)
Collaborators: CHI St. Luke's Health, Texas (Other); Aldagen (Industry)
Responsible Party: Principal Investigator, Emerson Perin, MD, PhD, Director Clinical Research for Cardiovascular Medicine and Stem Cell Center, Texas Heart Institute
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: UT-H-GEN-05-0599
Record Dates: First submitted 2006-04-10; First posted 2006-04-13 (Estimated); Results first posted 2015-11-23 (Estimated); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Coronary Artery Disease
Keywords: stem cell; autologous; ischemia
MeSH Terms: conditions — Coronary Artery Disease; Ischemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stem Cell Therapy (Active Comparator): Subjects are randomized to receive Stem Cell Therapy (treatment) at the time of enrollment where cells are delivered after NOGA mapping and cells injected with the Myostar catheter.
  Interventions: Biological: Stem Cell Therapy
- Control (Placebo Comparator): Placebo patients will receive injections of plasma (control) instead of stem cells. Placebo patients are able to crossover and receive active treatment at 6 months if they meet the criteria.
  At 6 months, subject is offered stem cell therapy and then followed for 12 months.
  Interventions: Other: Control (plasma)

INTERVENTIONS:
Biological: Stem Cell Therapy — Cells are injected under electromechanical guidance and delivered by the Myostar catheter after NOGA mapping.
  Other Names: NOGA Myostar catheter
  Arms: Stem Cell Therapy
Other: Control (plasma) — Placebo patients receive an injection of plasma (control) containing 5 % albumin the the same quantity as the stem cell arm. A total of 15 injections of 0.2 ml to total 3.0 ml.
  Arms: Control

SUMMARY:
Recent studies have suggested that it may be possible to grow new blood vessels (angiogenesis) to supply the heart muscle that is currently not getting enough blood. One theory is that a certain type of stem cell, aldehyde dehydrogenase bright stem cells, may stimulate the growth of new vessels. After a bone marrow procedure, the special cells are separated and then injected back into the heart around the area of damage with a special guidance and injection system.

Once a patient meets all inclusion criteria and no exclusion criteria, he/she will be consented to the study and extensive baseline testing will be completed at St. Luke's Episcopal Hospital in Houston, Texas. Once all baseline criteria are met, the patient has his/her own bone marrow harvested and later injected, if randomized to receive active treatment. The day after the bone marrow harvest, the patient is taken to the cardiac catheterization lab where NOGA mapping is performed and the processed cells or placebo are injected under electromechanical guidance into the affected areas of the left ventricle. The patient is usually discharged home the next day and returns for follow-up at weeks 1 and 4, and months 3 and 6, and at one year unless there is a crossover and then he/she begins baseline again at 6 months and follow-up for one more year. Follow-up testing, including quality of life and NOGA mapping, is done at the time of injection, as well as at 6 months.

DETAILED DESCRIPTION:
This is a phase I, double blind trial to evaluate the use of Aldehyde Dehydrogenase-Bright (ALDHbr) in ischemic cardiomyopathy patients. The study hypothesis is that transendocardial injections of autologous bone marrow cells in patients with end-stage ischemic heart disease is safe, can provide neovascularization, and can improve perfusion and myocardial contractility. The primary object of this study is to assess the safety of the ALDHbr cell injections. The efficacy will be based upon treadmill MVO2. A maximum of 60 patients will be enrolled in the study. At the end of 6 months, after the required testing has been completed, the patients will be told whether they were in the control group or not. The patients in the control group will be given the option to crossover and actually receive stem cell injection. At the time of crossover, which then becomes the baseline, patients will begin the follow-up with all testing including clinic visits for one year for a total of 18 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Canadian cardiovascular (CV) Class II-IV angina and/or congestive heart failure (CHF) symptoms
* Ejection fraction less than or equal to 45%
* Reversible perfusion defect on single photon emission computed tomography (SPECT)
* Coronary artery disease (CAD) unable to be corrected by surgery (bypass) or intervention (stent)
* Able to walk on treadmill
* Hemodynamically stable

Exclusion Criteria:

* Age less than 18 or greater than 70
* Atrial fibrillation
* Severe valve disease
* History of cancer in last 5 years
* HIV positive; hepatitis B or C positive.
* Left ventricular wall thickness less than 8 mm
* Recent heart attack within the last 30 days

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2006-04; Primary Completion 2009-08 (Actual); Study Completion 2023-08-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emerson Perin, MD, PhD, Principal Investigator — Texas Heart Institute
Locations (1):
- Texas Heart Institute/Baylor St. Luke's Medical Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Relevant results are summarized and published. No need for individual results to be shared.

REFERENCES:
- [Background] Perin EC, Silva GV, Zheng Y, Gahremanpour A, Canales J, Patel D, Fernandes MR, Keller LH, Quan X, Coulter SA, Moore WH, Herlihy JP, Willerson JT. Randomized, double-blind pilot study of transendocardial injection of autologous aldehyde dehydrogenase-bright stem cells in patients with ischemic heart failure. Am Heart J. 2012 Mar;163(3):415-21, 421.e1. doi: 10.1016/j.ahj.2011.11.020. Epub 2012 Feb 10. PMID 22424012
- See also: The link is to Texas Heart Institute's Stem Cell Department home page. — http://www.texasheart.org/stemcell

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twenty one patients were recruited between 9/1/06 and 8/6/08 from outpatient Cardiology clinics.
Groups:
- Control: Placebo patients will receive injections of plasma (control) instead of stem cells. Placebo patients are able to crossover and receive active treatment at 6 months if they meet the criteria.
  Plasma control: Placebo patients receive an injection of plasma containing 5 % albumin the the same quantity as the stem cell arm. A total of 15 injections of 0.2 ml to total 3.0 ml.
Period: Overall Study
Arm/Group | Stem Cell Therapy | Control
Started | 11 | 10
Completed | 10 | 10
Not Completed | 1 | 0
Not completed — not treated due to patient medical condi | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Control: Control (Placebo) patients will receive injections of plasma control instead of stem cells. Placebo patients are able to crossover and receive active treatment at 6 months if they meet the criteria.
  Plasma control: Placebo patients receive an injection of plasma containing 5 % albumin the the same quantity as the stem cell arm. A total of 15 injections of 0.2 ml to total 3.0 ml.
- Total: Total of all reporting groups
Arm/Group | Stem Cell Therapy | Control | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 20
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age | 58.2 (6.1) | 57.8 (5.5) | 58.0 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 9 | 8 | 17
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Safety of Aldehyde Dehydrogenase Bright Stem Cells Versus the Control Group as Measured by Combined Early and Late Adverse Events
Description: Safety of cell injections was assessed by reviewing adverse events at 2 time points: Baseline (periprocedural period up to 2 weeks post-procedure) and at 6 months post-procedure. Major adverse events were adjudicated (hospitalization, arrhythmia, exacerbation of congestive HF [CHF], acute coronary syndrome, myocardial infarction, stroke, or death).
Time Frame: Baseline and 6 months
Population: The data was analyzed for all participants in control and treated groups.
Measure: Number; unit: participants
Groups:
- Control: Placebo patients will receive injections of plasma (control) instead of stem cells. Placebo patients are able to crossover and receive active treatment at 6 months if they meet the criteria.
  At 6 months, subject is offered stem cell therapy and then followed for 12 months.
  Control (plasma): Placebo patients receive an injection of plasma (control) containing 5 % albumin the the same quantity as the stem cell arm. A total of 15 injections of 0.2 ml to total 3.0 ml.
- Stem Cell Therapy: Subject is randomized to receive intramyocardial injection of stem cells (stem cell therapy) via NOGA mapping.
Arm/Group | Control | Stem Cell Therapy
Number analyzed (Participants) | 10 | 10
participants
  Number treated | 10 | 10
  atrial arrhythmia | 0 | 2
  EMM realted ventricular tachycardia | 2 | 0
  EMM related ventricular fibrillation | 1 | 0
  cerebrovascular event | 1 | 0
  angina exacerbation | 1 | 5
  myocardial infarction (NSTEMI) | 0 | 1
  intracardiac thrombus | 0 | 1

2. Secondary Outcome: New York Heart Association (NYHA) Classification
Description: Clinical and functional assessment in endstage ischemic cardiomyopathy patients using New York Heart Association (NYHA)Classification and indicates extent of heart failure based on limitations in physical activity.
  Class I- No symptoms/limitation in ordinary physical activity (shortness of breath when walking, etc) Class II-Mild symptoms/slight limitation during ordinary activity Class III- Marked limitation in activity due to symptoms, even during less-than-ordinary activity Class IV- Severe limitations in activity/experiences symptoms while at rest (bedbound)
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: NYHA Functional class
Arm/Group | Stem Cell Therapy | Control
Number analyzed (Participants) | 10 | 10
NYHA Functional class
  NYHA baseline | 2.5 (0.5) | 2.6 (0.5)
  NYHA 6 months | 2.3 (0.5) | 2.1 (0.3)

3. Secondary Outcome: Canadian Cardiovascular (CCS) Angina Score
Description: Clinical and functional assessment in endstage ischemic cardiomyopathy patients using Canadian Cardiovascular (CCS) Angina Score which indicates discomfort from angina (chest pain).
  Class I- Angina only during strenuous or prolonged activity Class II- Slight limitation, with angina only during vigorous physical activity Class III- Symptoms with everyday living activities (moderate limitation) Class IV- Inability to perform any activity without angina or angina at rest (severe limitation)
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stem Cell Therapy | Control
Number analyzed (Participants) | 10 | 10
units on a scale
  CCS baseline | 2.5 (0.5) | 2.5 (0.5)
  CCS 6 months | 2.0 (0.0) | 2.0 (0.5)

4. Secondary Outcome: Echocardiography (EF)Percent (%)
Description: Clinical and functional assessment in endstage ischemic cardiomyopathy patients using Echocardiography measures ejection fraction(EF)as a percentage(%) of blood leaving the heart with each beat or contraction. It can provide information concerning structural characteristics and blood flow in the heart and blood vessels. A normal heart pumps 50-75% of the blood with each contraction.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: percentage of blood
Arm/Group | Stem Cell Therapy | Control
Number analyzed (Participants) | 10 | 10
percentage of blood
  baseline | 36.1 (10.9) | 32.1 (10.6)
  6 months | 36.0 (11.3) | 34.0 (9.3)

5. Secondary Outcome: Left Ventricular End-Systolic Volume (LVESV) (ml)
Description: Clinical and functional assessment in endstage ischemic cardiomyopathy patients using Left Ventricular End-Systolic Volume (LVESV) when the blood moves from the ventricles to the atria during the contraction cycle. Measured as volume in milliliters (ml). Normal is approximately 60- 65 milliliters.
Time Frame: baseline and 6 months
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Stem Cell Therapy | Control
Number analyzed (Participants) | 10 | 9
ml
  LVESV baseline | 93.2 (46.1) | 94.9 (59.8)
  LVESV 6 months | 85.9 (46.2) | 94.7 (62.2)

6. Secondary Outcome: Left Ventricular End-Diastolic Volume (LVEDV)
Description: Clinical and functional assessment in endstage ischemic cardiomyopathy patients using Left Ventricular End-Diastolic Volume (LVEDV)which is the volume of blood inside the left ventricle when the heart has completed its filling cycle. The volume of the left ventricle is measured during contraction and relaxation. Normal heart volume inside the left ventricle is about 140 milliliters.
Time Frame: baseline and 6 months
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Stem Cell Therapy | Control
Number analyzed (Participants) | 10 | 10
ml
  LVDEV baseline | 138.3 (43.0) | 132.7 (65.2)
  LVDED 6 months | 127.2 (51.3) | 131.3 (67.4)

7. Secondary Outcome: Echocardiography Wall Motion Score Index (WMSI)
Description: Clinical and functional assessment in endstage ischemic cardiomyopathy patients using Echocardiography Wall Motion Score Index (WMSI) as defined by the American Heart Association which allows detection of abnormalities in the heart wall or blood flowing through the heart. Using this model, the left ventricle is divided into 17 segments. Normal contracting Left Ventricle has WMSI of 1. Larger WMSI indicates higher degree of abnormalities (2 for hypokinetic, 3 for akinetic, 4 for dyskinetic, and 5 for aneurysmal). WMSI was calculated as the sum of scores divided by the total number of segments.
Time Frame: baseline and 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stem Cell Therapy | Control
Number analyzed (Participants) | 10 | 10
units on a scale
  WMSI baseline | 1.91 (0.51) | 2.13 (0.38)
  WMSI 6 months | 1.90 (0.57) | 2.06 (0.41)

8. Secondary Outcome: Myocardial Oxygen Consumption (MVO2)
Description: Clinical and functional assessment in endstage ischemic cardiomyopathy patients using Myocardial Oxygen Consumption (MVO2)which is the amount of oxygen used by the heart muscle and is indicative of heart muscle function. Normal value is 15.5 Volume %. Measured as milliliters (ml) oxygen per kilogram (kg) body weight per minute.
Time Frame: baseline and 6 months
Population: data from 9 stem cell patients at 6 months, 10 at baseline
Measure: Mean (Standard Deviation); unit: ml/kg/min
Arm/Group | Stem Cell Therapy | Control
Number analyzed (Participants) | 10 | 9
ml/kg/min
  MVO2 baseline | 15.5 (6.3) | 14.1 (4.8)
  MVO2 6 months | 17.7 (4.1) | 14.6 (6.7)

9. Secondary Outcome: Echocardiography (EF) Percent (%)
Description: as for outcome 4
Time Frame: baseline and 6 months
Measure: Mean (Standard Deviation); unit: percentage of blood
Arm/Group | Stem Cell Therapy | Control
Number analyzed (Participants) | 8 | 7
percentage of blood
  EF (%) baseline | 38.0 (17.5) | 41.9 (11.8)
  EF (%) 6 months | 40.4 (15.8) | 42.2 (7.6)

10. Secondary Outcome: Total Severity Score (Stress)
Description: For the stress test, cardiac SPECT polar mapping (gated dual-isotope) is used to evaluate perfusion, compared against a database with a statistically significant number of polar maps of healthy hearts based on gender, data acquisition method, stress vs rest and type of data (i.e. perfusion, wall motion or wall thickening) using a clinically validated software package (J Nucl Med Technol 2006; 34:3-17). The basal and mid-ventricle heart wall is mapped by cylindrical sampling and apex mapped by spheric, cylindric and radial sampling.
  Total severity score during stress is the sum of blackout pixels in the blackout polar map of myocardial perfusion during stress using cardiac SPECT imaging (adding scores in different views), weighted by the number of SDs below the mean.
  Total severity score varies from 0 (normal) to several thousands although the upper limit is not well defined. A score greater than 1000 indicates poor perfusion.
Time Frame: baseline and 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stem Cell Therapy | Control
Number analyzed (Participants) | 10 | 10
units on a scale
  Stress Severity Score (stress) baseline | 798.2 (528.7) | 1007.6 (352.4)
  Stress Severity Score (stress) 6 months | 785.9 (554.6) | 1132 (588.5)

11. Secondary Outcome: Total Severity Score (Rest)
Description: For the total severity score at rest, cardiac SPECT polar mapping (gated dual-isotope) is used to evaluate myocardial cardiac perfusion, compared against a database with a statistically significant number of polar maps of healthy hearts and compared based on gender, data acquisition method, stress vs rest and type of data (i.e. perfusion, wall motion or wall thickening) using a clinically validated software package (J Nucl Med Technol 2006; 34:3-17). The basal and mid-ventricle heart wall is mapped by cylindrical sampling and apex mapped by spheric, cylindric and radial sampling at rest.
  Total severity score at rest is the sum of blackout pixels in the rest blackout polar map of myocardial perfusion cardiac SPECT imaging (adding scores in different views), weighted by the number of SDs below the mean.
  Total severity score varies from 0 (normal) to several thousands although the upper limit is not well defined. A score greater than 1000 indicates poor perfusion.
Time Frame: baseline and 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stem Cell Therapy | Control
Number analyzed (Participants) | 10 | 10
units on a scale
  Total Severity Score (rest) baseline | 542.8 (440.7) | 812.4 (304.5)
  Total Severity Score (rest) 6 months | 594.6 (488.9) | 828 (396.9)

12. Secondary Outcome: Total Severity Score (Reversible)
Description: For the severity test, cardiac SPECT polar mapping (gated dual-isotope) is used to evaluate myocardial cardiac perfusion, compared against a database with a statistically significant number of polar maps of healthy hearts and compared based on gender, data acquisition method, stress vs rest and type of data (i.e. perfusion, wall motion or wall thickening) using clinically validated software package (J Nucl Med Technol 2006; 34:3-17). The basal and mid-ventricle heart wall is mapped by cylindrical sampling and apex mapped by spheric, cylindric and radial sampling at rest/stress.
  Total severity score is the sum of blackout pixels in rest/stress blackout polar map of myocardial perfusion cardiac SPECT imaging (adding scores in different views), weighted by number of SDs below mean. Total severity score reversible is total severity scores at rest subtracted from those during stress. The severity score varies from 0 (normal) to > 1000 (poor perfusion) but upper limit is not well defined.
Time Frame: baseline and 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stem Cell Therapy | Control
Number analyzed (Participants) | 10 | 10
units on a scale
  Total Severity Score (reversible) baseline | 72.6 (95.2) | 46.5 (48.5)
  Total Severity Score (reversible) 6 months | 22.9 (39.2) | 87.3 (60.2)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected pre-procedure, during procedure, after procedure, week 1, week 4, month 3 and month 6 post-procedure.
Groups:
- Control: Placebo (control) patients will receive injections of plasma control instead of stem cells. Placebo patients are able to crossover and receive active treatment at 6 months if they meet the criteria.
  Plasma control: Placebo patients receive an injection of plasma containing 5 % albumin the the same quantity as the stem cell arm. A total of 15 injections of 0.2 ml to total 3.0 ml.
Arm/Group | Stem Cell Therapy | Control
Serious Adverse Events (participants affected / at risk) | 10/10 | 10/10
Other Adverse Events (participants affected / at risk) | 10/10 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stem Cell Therapy (N=10) | Control (N=10)
non-ST elevation MI/acute non-ST elevation MI (Cardiac disorders) | 1 (1) | 2 (2)
ventricular tachycardia /ventricular tachycardia (ICD shocks)/ ventricular arrhythmia (Cardiac disorders) | 2 (2) | 2 (2)
new stenotic lesion in SVG to RCA (Cardiac disorders) | 1 (1) | 0 (0)
acute congestive heart failure (Cardiac disorders) | 0 (0) | 1 (1)
inappropriate AICD function (Cardiac disorders) | 1 (1) | 0 (0)
bilateral eye cataracts (Eye disorders) | 1 (1) | 0 (0)
left eye macular edema (Eye disorders) | 1 (1) | 0 (0)
lightheadness or dizziness (General disorders) | 2 (2) | 0 (0)
cholelithiasis (Gastrointestinal disorders) | 0 (0) | 1 (1)
postoperative hematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fentanyl overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
mild bleeding at right groin cath site (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
intracerebral hemorrhage/ ischemic stroke/ embolic stroke (Nervous system disorders) | 1 (1) | 2 (2)
increased shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
community acquired pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
increased claudication (Vascular disorders) | 1 (1) | 0 (0)
dehydration (General disorders) | 0 (0) | 1 (1)
fever of unknown origin (General disorders) | 0 (0) | 1 (1)
hospitalization for sinusitis (Infections and infestations) | 0 (0) | 1 (1)
hypotension (Cardiac disorders) | 0 (0) | 1 (1)
ideoventricular rhythm (Cardiac disorders) | 0 (0) | 1 (1)
ischemic cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stem Cell Therapy (N=10) | Control (N=10)
second degree AV block, type 2 (Cardiac disorders) | 1 (1) | 0 (0)
acute bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
acute renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
altered mental status (Psychiatric disorders) | 1 (1) | 0 (0)
decreased platelet count (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
irregular heart rhythm (Cardiac disorders) | 0 (0) | 1 (1)
left ventricular thrombus (Cardiac disorders) | 0 (0) | 1 (1)
hypotension (Cardiac disorders) | 2 (3) | 3 (4)
increased troponin level (Cardiac disorders) | 1 (1) | 0 (0)
increased cardiac chest pain (Cardiac disorders) | 4 (4) | 1 (1)
atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
exacerbation of congestive heart failure (Cardiac disorders) | 0 (0) | 4 (4)
heart racing (Cardiac disorders) | 0 (0) | 2 (2)
hypertension elevation (Cardiac disorders) | 1 (1) | 0 (0)
new onset of atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
increased CPK (Cardiac disorders) | 0 (0) | 1 (1)
chest pain- nonspecific (Cardiac disorders) | 0 (0) | 1 (1)
possible apical thrombus (Cardiac disorders) | 0 (0) | 1 (1)
episode of atypical cardiac chest pain (Cardiac disorders) | 1 (2) | 0 (0)
left ventricular apical thrombus (Cardiac disorders) | 1 (1) | 0 (0)
sustained ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
diaphoresis (Cardiac disorders) | 0 (0) | 1 (1)
short periods of atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
labyrinthitis (Ear and labyrinth disorders) | 0 (0) | 1 (1)
increased hearing loss (Ear and labyrinth disorders) | 0 (0) | 1 (1)
elevated blood glucose (Endocrine disorders) | 0 (0) | 1 (2)
low testosterone level (Endocrine disorders) | 0 (0) | 1 (1)
photophobia (Eye disorders) | 0 (0) | 1 (1)
stomach flu (Gastrointestinal disorders) | 1 (1) | 0 (0)
vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0)
rectal polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
worsening constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
epigastric pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
fatigue (General disorders) | 3 (4) | 5 (7)
cold symptoms (General disorders) | 0 (0) | 1 (1)
nasal discharge (General disorders) | 1 (1) | 0 (0)
productive cough (General disorders) | 1 (1) | 0 (0)
fever (General disorders) | 2 (2) | 2 (2)
obstructive sleep apnea (General disorders) | 0 (0) | 1 (1)
headache (General disorders) | 2 (2) | 1 (1)
TIA symptoms (General disorders) | 0 (0) | 1 (1)
cough (General disorders) | 1 (1) | 0 (0)
drowsiness (General disorders) | 1 (1) | 0 (0)
nausea (General disorders) | 1 (1) | 2 (3)
syncope (General disorders) | 1 (1) | 0 (0)
weight loss (General disorders) | 1 (1) | 1 (1)
bleeding from bone marrow site (General disorders) | 0 (0) | 1 (1)
vertigo (General disorders) | 0 (0) | 1 (1)
intermittent right frontal headache (General disorders) | 0 (0) | 1 (1)
dehydration (General disorders) | 0 (0) | 1 (1)
dizziness, lightheadedness (General disorders) | 2 (2) | 4 (4)
weight gain (General disorders) | 1 (1) | 0 (0)
abnormal sleep pattern (General disorders) | 0 (0) | 1 (1)
nasal congestion (General disorders) | 0 (0) | 2 (3)
athlete's foot (General disorders) | 0 (0) | 1 (1)
lower extremity edema (General disorders) | 0 (0) | 2 (3)
bodyache (General disorders) | 0 (0) | 1 (1)
chills (General disorders) | 0 (0) | 1 (1)
poison oak exposure (General disorders) | 0 (0) | 1 (1)
rash (General disorders) | 0 (0) | 1 (1)
Bells Palsey (General disorders) | 0 (0) | 1 (1)
rash to neck and upper chest (General disorders) | 0 (0) | 1 (1)
rash from Holter (General disorders) | 0 (0) | 1 (1)
nose bleed (General disorders) | 0 (0) | 1 (1)
tooth decay (General disorders) | 0 (0) | 1 (1)
difficulty maintaining sleep (General disorders) | 1 (1) | 0 (0)
forgetfullness (General disorders) | 1 (1) | 0 (0)
mild headache after 6 min walk (General disorders) | 1 (1) | 0 (0)
bruised forehead due to fall (General disorders) | 1 (1) | 0 (0)
minor burns (from Halter electrodes) (General disorders) | 0 (0) | 1 (1)
flu-like syndrome (General disorders) | 0 (0) | 1 (1)
cold feet (General disorders) | 1 (1) | 0 (0)
facial numbness (General disorders) | 1 (1) | 0 (0)
numbness in extremity (General disorders) | 1 (1) | 0 (0)
increased liver function tests (Hepatobiliary disorders) | 0 (0) | 1 (1)
leukocytosis (Immune system disorders) | 1 (1) | 0 (0)
sinus infection (Infections and infestations) | 5 (6) | 3 (3)
strep throat (Infections and infestations) | 1 (1) | 0 (0)
viral syndrome (Infections and infestations) | 1 (1) | 0 (0)
Herpes Simplex (Infections and infestations) | 0 (0) | 1 (1)
influenza (Infections and infestations) | 1 (1) | 1 (1)
tooth infection (Infections and infestations) | 0 (0) | 1 (1)
infection of right index finger (Infections and infestations) | 1 (1) | 0 (0)
pain at bone marrow harvest site (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
hypoglycemic (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
fluctuating glucose (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
symptomatic volume depletion (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
cervial neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
bilateral knee pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
pain in left arm (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
left leg cramps (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
left chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
bone spurs in neck and spine (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
chipped bone fragment in neck (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
bulging disk at lower back (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
injured miniscus (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
bilateral thigh pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
soreness in feet (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
left foot fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
sore left arm (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
sore left knee (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
back tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
increase of chronic back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
shoulder pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
bilateral hyperreflexia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
anxiety (Psychiatric disorders) | 0 (0) | 2 (2)
increased forgetfulness (Psychiatric disorders) | 0 (0) | 1 (1)
psychological stress (Psychiatric disorders) | 1 (1) | 0 (0)
urinary tract infection (Renal and urinary disorders) | 0 (0) | 1 (1)
elevated blood urea nitrogen (BUN) (Renal and urinary disorders) | 0 (0) | 1 (1)
elevated creatinine level (Renal and urinary disorders) | 0 (0) | 1 (1)
exacerbation of preexisting disease- kidney stones (Renal and urinary disorders) | 0 (0) | 1 (1)
renal insufficiency (Renal and urinary disorders) | 0 (0) | 1 (1)
large right renal cyst (Renal and urinary disorders) | 1 (1) | 0 (0)
atrophic vaginitis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1)
increased shortness of breath (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1)
non-productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
chest congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
plantar fascitis (Vascular disorders) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
The study is a preliminary study based on a small sample size which limits the statistical rigor of the analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes